CLINICAL TRIAL: NCT01826916
Title: EDEMA2: An Open-Label Study to Assess the Efficacy and Tolerability of Repeated Doses of DX-88 (Recombinant Plasma Kallikrein Inhibitor) in Patients With Hereditary Angioedema
Brief Title: EDEMA2: Evaluation of DX-88's Effect in Mitigating Angioedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DX-88/5; EDEMA2 (Other: Dyax)
Record Dates: First submitted 2012-02-16; First posted 2013-04-09 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — ecallantide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 5mg/m2 DX-88 IV (Experimental): 5mg/m2 DX-88 (ecallantide)administered intravenously
  Interventions: Drug: DX-88 (ecallantide)
- 10mg/m2 DX-88 IV (Experimental): 10mg/m2 DX-88(ecallantide)administered intravenously
  Interventions: Drug: DX-88 (ecallantide)
- 20mg/m2 DX-88 IV (Experimental): 20mg/m2 DX-88 (ecallantide) administered intravenously
  Interventions: Drug: DX-88 (ecallantide)
- 30 mg DX-88 SC (Experimental): 30mg DX-88(ecallantide)administered subcutaneously
  Interventions: Drug: DX-88 (ecallantide)

INTERVENTIONS:
Drug: DX-88 (ecallantide) — solution for injection 10 mg/mL

SUMMARY:
EDEMA2 is an open-label, Phase 2 dose-ranging study designed to assess the safety and efficacy of repeated dosing of DX-88 (recombinant plasma kallikrein inhibitor) in Patients with Hereditary Angioedema.

ELIGIBILITY:
Inclusion Criteria:

* 10 years of age or older
* Documented diagnosis of HAE (Type I or II)
* Patient reported to a study site no later than 4 hours following patient recognition of the onset of the attack
* Willing and able to give informed consent

Exclusion Criteria:

* Patients with a serious intercurrent illness or serious active infection
* Patient with serum creatinine greater than 110% the upper limit of normal or liver transaminases 2 times the upper limit of normal
* Receipt of an investigational drug or device, within 30 days prior to study treatment
* Pregnancy or breastfeeding
* Diagnosis of acquired angioedema (AAE)
* Patients who had not completed their Day-7 follow-up procedures for a previously treated attack

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-11-01 (Actual); Primary Completion 2005-12-01 (Actual); Study Completion 2006-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of attacks treated with successful outcome | 24 hours
  successful outcome is defined as attack resolution begun within 4 hrs after treatment and maintained for 24 hours
Proportion of attacks with a partial response | 24 hours
  partial response is defined as an initial response to dosing followed by a relapse within 4 to 24 hours

SECONDARY OUTCOMES:
Proportion of patients who respond to a 2nd dose of ecallantide after an initial, partial response | 24 hours
Time to resolution onset of each acute attack, as determined by patient report | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Derived] Rubinstein E, Stolz LE, Sheffer AL, Stevens C, Bousvaros A. Abdominal attacks and treatment in hereditary angioedema with C1-inhibitor deficiency. BMC Gastroenterol. 2014 Apr 9;14:71. doi: 10.1186/1471-230X-14-71. PMID 24712435
- [Derived] MacGinnitie AJ, Davis-Lorton M, Stolz LE, Tachdjian R. Use of ecallantide in pediatric hereditary angioedema. Pediatrics. 2013 Aug;132(2):e490-7. doi: 10.1542/peds.2013-0646. Epub 2013 Jul 22. PMID 23878046